CLINICAL TRIAL: NCT02742103
Title: A Phase 2, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group, Study to Investigate the Safety and Tolerability of Multiple Dose Administration of CSL112 in Subjects With Moderate Renal Impairment and Acute Myocardial Infarction
Brief Title: A Study of CSL112 in Adults With Moderate Renal Impairment and Acute Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CSL112_2001; 2015-003017-26 (EudraCT Number)
Record Dates: First submitted 2016-03-30; First posted 2016-04-18 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Acute Myocardial Infarction; Moderate Renal Impairment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CSL_112 (Experimental): CSL112 will be administered intravenously, once weekly for 4 consecutive weeks (4 infusions in total).
  Interventions: Biological: CSL_112
- Placebo (Placebo Comparator): Placebo will be administered at the same frequency, volume and duration as the CSL112 infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CSL_112 — CSL112 is a novel formulation of apolipoprotein A-I (apoA-I) purified from human plasma and reconstituted to form high-density lipoprotein (HDL) particles.
  Arms: CSL_112
Other: Placebo — 0.9% weight/volume sodium chloride solution (ie, normal saline)
  Arms: Placebo

SUMMARY:
This study is a phase 2, multicenter, double-blind, randomized, placebo controlled, parallel-group study to investigate the renal safety and tolerability of multiple dose intravenous (IV) administration of CSL112 compared with placebo in subjects with moderate renal impairment (RI) and acute myocardial infarction (AMI).

ELIGIBILITY:
Inclusion Criteria:

• Men or women, at least 18 years of age, with evidence of moderate renal impairment (an eGFR ≥ 30 and <60 mL/min/1.73 m2) and myocardial necrosis in a clinical setting consistent with a type I (spontaneous) acute myocardial infarction (AMI).

Exclusion Criteria:

* Symptoms, biomarker elevation or electrocardiogram (ECG) changes other than those of the index event that are consistent with a diagnosis of AMI but are likely not due to primary myocardial ischemia
* Ongoing hemodynamic instability
* Planned coronary artery bypass surgery
* Evidence of hepatobiliary disease
* History of acute kidney injury (AKI) after previous exposure to an intravenous contrast agent.
* History of nephrotic range proteinuria.
* Known history of allergy to soy beans or peanuts, immunoglobulin A (IgA) deficiency, antibodies to IgA , or hypersensitivity to CSL112 or any of its components.
* Other severe comorbid condition, concurrent medication, or other issue that renders the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Duffy, MD, Study Director — CSL Behring
Locations (31):
- United States (13):
  - Study Site 16101, Birmingham, Alabama
  - Study Site 16078, Huntsville, Alabama
  - Study Site 16168, Concord, California
  - Study Site 16130, Littleton, Colorado
  - Study Site 16135, Danbury, Connecticut
  - Study Site 16003, Jacksonville, Florida
  - Study Site 16112, Boise, Idaho
  - Study Site 16208, Alexandria, Louisiana
  - Study Site 16061, Petoskey, Michigan
  - Study Site 16056, Durham, North Carolina
  - Study Site 16014, High Point, North Carolina
  - Study Site 16018, Rapid City, South Dakota
  - Study Site 16241, Wichita Falls, Texas
- Germany (6):
  - Study Site 17001, Freiburg im Breisgau, Baden-Wurttemberg
  - Study Site 17014, Frankfurt am Main, Hesse
  - Study Site 17005, Berlin
  - Study Site 17009, Berlin
  - Study Site 17003, Berlin
  - Study Site 17006, Hamburg
- Hungary (5):
  - Study Site 18001, Budapest
  - Study Site 18005, Budapest
  - Study Site 18007, Nyíregyháza
  - Study Site 18003, Pécs
  - Study Site 18009, Szeged
- Israel (3):
  - Study Site 19005, Haifa
  - Study Site 19002, Nahariya
  - Study Site 19008, Safed
- Netherlands (4):
  - Study Site 21001, Alkmaar
  - Study Site 21006, Amsterdam
  - Study Site 21017, Amsterfoort
  - Study Site 21008, Nijmegen

REFERENCES:
- [Derived] Zheng B, Duffy D, Tricoci P, Kastrissios H, Pfister M, Wright SD, Gille A, Tortorici MA. Pharmacometric analyses to characterize the effect of CSL112 on apolipoprotein A-I and cholesterol efflux capacity in acute myocardial infarction patients. Br J Clin Pharmacol. 2021 Jun;87(6):2558-2571. doi: 10.1111/bcp.14666. Epub 2020 Dec 23. PMID 33217027
- [Derived] Gibson CM, Kerneis M, Yee MK, Daaboul Y, Korjian S, Mehr AP, Tricoci P, Alexander JH, Kastelein JJP, Mehran R, Bode C, Lewis BS, Mehta R, Duffy D, Feaster J, Halabi M, Angiolillo DJ, Duerschmied D, Ophuis TO, Merkely B. The CSL112-2001 trial: Safety and tolerability of multiple doses of CSL112 (apolipoprotein A-I [human]), an intravenous formulation of plasma-derived apolipoprotein A-I, among subjects with moderate renal impairment after acute myocardial infarction. Am Heart J. 2019 Feb;208:81-90. doi: 10.1016/j.ahj.2018.11.008. Epub 2018 Nov 22. PMID 30580130

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: To ensure that at least 1/3 of the study population had an estimated glomerular filtration (eGFR) in the chronic kidney disease (CKD) Stage 3b range, no more than 2/3 of the study population were to have an eGFR in the CKD Stage 3a range. Randomization was stratified by eGFR and by medical history of diabetes.
Period: Overall Study
Arm/Group | CSL_112 | Placebo
Started | 55 | 28
Completed | 46 | 23
Not Completed | 9 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Moved to another town | 0 | 1
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSL_112 | Placebo | Total
Number analyzed (Participants) | 55 | 28 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (10.95) | 71.9 (10.12) | 71.1 (10.63)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 11 | 4 | 15
  65-84 years | 42 | 23 | 65
  85 years and over | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 37 | 18 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 52 | 28 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 8 | 2 | 10
  Hungary | 20 | 8 | 28
  United States | 10 | 9 | 19
  Israel | 5 | 5 | 10
  Germany | 12 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With at Least One Occurrence of Treatment-emergent Renal Serious Adverse Events (SAEs) (SAF)
Description: A renal SAE is defined as any SAE with a MedDRA preferred term included in the Acute Renal Failure narrow Standard MedDRA Query or a preferred term of renal tubular necrosis, renal cortical necrosis, renal necrosis, or renal papillary necrosis.
Time Frame: Up to 9 weeks
Population: The Safety (SAF) Population consisted of all subjects who received at least a partial dose of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
percentage of participants | 1.9 | 14.3
Statistical Analysis 1: Comparison: CSL_112 vs Placebo; Test type: Other; Newcombe-Wilson; Rate difference (CSL112 - placebo) = -0.124, 95% CI 2-sided [-0.296 to -0.005]

2. Primary Outcome: Percent of Participants With Treatment-emergent Acute Kidney Injury (AKI )
Description: Acute kidney injury is defined as an absolute increase in serum creatinine from baseline ≥ 0.3 mg/dL during the Active Treatment Period that is sustained upon repeat measurement by the central laboratory no earlier than 24 hours after the elevated value. If no repeat value is obtained, a single serum creatinine value that is increased from baseline ≥ 0.3 mg/dL (26.5 μmol/L) during the Active Treatment Period would also fulfil the definition of AKI.
Time Frame: Up to 4 weeks
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 50 | 28
percentage of participants | 4.0 | 14.3
Statistical Analysis 1: Comparison: CSL_112 vs Placebo; Test type: Other; Newcombe-Wilson; Rate difference (CSL112 - placebo) = -0.103, 95% CI 2-sided [-0.277 to 0.025]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Time Frame: Up to 9 weeks
Population: SAF
Measure: Number; unit: participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
participants | 38 | 20

4. Secondary Outcome: Percentage of Participants With TEAEs
Time Frame: Up to 9 weeks
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
percentage of participants | 73.1 | 71.4

5. Secondary Outcome: Total Number of TEAEs
Time Frame: Up to 9 weeks
Population: SAF
Measure: Number; unit: Number of TEAEs
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
Number of TEAEs | 111 | 61

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Drug Reaction (ADR) or Suspected ADR
Description: Adverse drug reactions or suspected adverse drug reactions are defined as:
  1. All TEAEs, including local tolerability events, that begin during or within 1 hour after the end of an infusion; or
  2. Those TEAEs that the investigator or sponsor indicate may be causally related to product administration; or
  3. All TEAEs for which the Investigator's causality assessment is missing or indeterminate; or
  4. All TEAEs for which the incidence in an active treatment arm exceeds the exposure-adjusted incidence rate in the placebo arm by 30% or more, provided the difference in incidence rates is 1% or more.
Time Frame: Up to 9 weeks
Population: SAF
Measure: Number; unit: participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
participants | 30 | 4

7. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Drug Reaction (ADR) or Suspected ADR
Description: as for outcome 6
Time Frame: Up to 9 weeks
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
percentage of participants | 57.7 | 14.3

8. Secondary Outcome: Number of Participants With Change in Renal Status
Description: Number of participants with changes in renal status defined as:
  * Absolute increases from baseline in serum creatinine as follows:
    i. ≤ baseline value ii. > 0 to < 0.3 mg/dL iii. ≥ 0.3 to ≤ 0.5 mg/dL iv. > 0.5 mg/dL
  * Increases in serum creatinine that are sustained for ≥ 24 hours upon repeat measurement that are greater than or equal to 1.5 x, 2 x, or 3.0 x the baseline value, or serum creatinine ≥ 4.0 mg/dL
  * Initiation of renal replacement therapy
  * Decrease in eGFR ≥ 25% from baseline starting during the active treatment period and that is sustained at the final study visit
Time Frame: Baseline and up to 4 weeks
Population: SAF
Measure: Number; unit: participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
participants
  ≤ baseline value | 9 | 3
  > 0 to < 0.3 mg/dL | 35 | 18
  ≥ 0.3 to ≤ 0.5 mg/dL | 4 | 4
  > 0.5 mg/dL | 2 | 2
  ≥ 1.5 × Baseline | 1 | 0
  ≥ 2 × Baseline | 0 | 0
  ≥ 3 × Baseline | 0 | 0
  ≥ 4.0 mg/dL | 0 | 0
  Decrease in eGFR by ≥ 25% | 5 | 4
  Initiation of renal replacement therapy | 0 | 1

9. Secondary Outcome: Percentage of Participants With Change in Renal Status
Description: Percentage of participants with changes in renal status defined as:
  * Absolute increases from baseline in serum creatinine as follows:
    i. ≤ baseline value ii. > 0 to < 0.3 mg/dL iii. ≥ 0.3 to ≤ 0.5 mg/dL iv. > 0.5 mg/dL
  * Increases in serum creatinine that are sustained for ≥ 24 hours upon repeat measurement that are greater than or equal to 1.5 x, 2 x, or 3.0 x the baseline value, or serum creatinine ≥ 4.0 mg/dL
  * Initiation of renal replacement therapy
  * Decrease in eGFR ≥ 25% from baseline starting during the active treatment period and that is sustained at the final study visit
Time Frame: Baseline and up to 4 weeks
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
percentage of participants
  ≤ Baseline Value | 17.3 | 10.7
  > 0 to < 0.3 mg/dL | 67.3 | 64.3
  ≥ 0.3 to ≤ 0.5 mg/dL | 7.7 | 14.3
  > 0.5 mg/dL | 3.8 | 7.1
  ≥ 1.5 × Baseline | 1.9 | 0
  ≥ 2 × Baseline | 0 | 0
  ≥ 3 × Baseline | 0 | 0
  ≥ 4.0 mg/dL | 0 | 0
  Decrease in eGFR by ≥ 25% | 9.6 | 14.3
  Initiation of renal replacement therapy | 0 | 3.6

10. Secondary Outcome: Number of Participants With Change in Hepatic Status
Description: Number of participants with a change from baseline in hepatic status and that is sustained for ≥ 24 hours upon repeat measurement, defined as:
  1. Alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN)
  2. ALT > 5 x ULN
  3. ALT > 10 x ULN
  4. Serum total bilirubin > 1.5 x ULN
  5. Serum total bilirubin > 2 x ULN
  6. Possible Hy's law cases, as defined in the FDA Guidance for Industry: Drug-Induced Liver Injury: Premarketing Clinical Evaluation (July 2009).
Time Frame: Baseline and up to 4 weeks
Population: SAF
Measure: Number; unit: participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
participants
  total bilirubin > 1.5 x ULN | 4 | 1
  total bilirubin > 2 x ULN | 1 | 0
  ALT > 3 x ULN | 0 | 0
  ALT > 5 x ULN | 0 | 0
  ALT > 10 x ULN | 0 | 0
  Possible Hy's law cases | 0 | 0

11. Secondary Outcome: Percentage of Participants With Change in Hepatic Status
Description: Percentage of participants with a change from baseline in hepatic status and that is sustained for ≥ 24 hours upon repeat measurement, defined as:
  1. Alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN)
  2. ALT > 5 x ULN
  3. ALT > 10 x ULN
  4. Serum total bilirubin > 1.5 x ULN
  5. Serum total bilirubin > 2 x ULN
  6. Possible Hy's law cases, as defined in the FDA Guidance for Industry: Drug-Induced Liver Injury: Premarketing Clinical Evaluation (July 2009).
Time Frame: Baseline and up to 4 weeks
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
percentage of participants
  total bilirubin > 1.5 x ULN | 7.7 | 3.7
  total bilirubin > 2 x ULN | 1.9 | 0
  ALT > 3 x ULN | 0 | 0
  ALT > 5 x ULN | 0 | 0
  ALT > 10 x ULN | 0 | 0
  Possible Hy's law cases | 0 | 0

12. Secondary Outcome: Number of Participants With Treatment-emergent Bleeding Events
Description: Bleeding events are as defined by the Bleeding Academic Research Consortium (BARC) criteria (Mehran et al., 2011).
Time Frame: Up to 9 weeks
Population: SAF
Measure: Number; unit: participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
participants | 7 | 5

13. Secondary Outcome: Percentage of Participants With Treatment-emergent Bleeding Events
Description: Bleeding events are as defined by the Bleeding Academic Research Consortium (BARC) criteria (Mehran et al., 2011).
Time Frame: Up to 9 weeks
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
percentage of participants | 13.5 | 17.9

14. Secondary Outcome: Percentage of Participants With Binding Antibodies Specific to Apolipoprotein A-I (Apo-A1) and CSL112
Time Frame: Up to 9 weeks
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
percentage of participants
  CSL112 antibody | 0 | 0
  apoA-I antibody | 0 | 0

15. Secondary Outcome: Baseline-corrected Plasma Concentration Maximum (Cmax) After Infusion 1 for apoA-I and PC
Time Frame: Immediately after end of infusion
Population: PK
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 52 | 28
mg/dL
  apoA-I | 124.6 (25.38) | -4.5 (9.46)
  PC | 198.4 (43.56) | -4.9 (15.04)

16. Secondary Outcome: Baseline-corrected Plasma Concentration Maximum (Cmax) After Infusion 4 for apoA-I and PC
Time Frame: Immediately after end of infusion
Population: PK
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL_112 | Placebo
Number analyzed (Participants) | 38 | 21
mg/dL
  apoA-I | 141.5 (41.11) | 1.4 (23.57)
  PC | 200.0 (71.78) | -13.2 (27.96)

17. Secondary Outcome: Plasma apoA-I and Phosphatidylcholine (PC) Accumulation Ratio After Infusion 4
Description: The plasma apoA-I and PC accumulation ratio will be determined for CSL112-treated subjects.
Time Frame: Immediately after end of infusion
Population: Pharmacokinetic Population (PK) consists of all subjects in the SAF who had at least 1 measurable plasma concentration of either apoA-I or PC.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CSL_112
Number analyzed (Participants) | 38
mg/dL
  apoA-I | 1.2 (0.32)
  PC | 1.0 (0.36)

ADVERSE EVENTS:
Time Frame: 67 days for each subject
Arm/Group | CSL_112 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/52 | 2/28
Serious Adverse Events (participants affected / at risk) | 12/52 | 10/28
Other Adverse Events (participants affected / at risk) | 18/52 | 12/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL_112 (N=52) | Placebo (N=28)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Gastrointestinal erosion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL_112 (N=52) | Placebo (N=28)
Hypertension (Vascular disorders) | 5 (5) | 1 (1)
Blood creatinine increased (Investigations) | 5 (5) | 0 (0)
Haemoglobin decreased (Investigations) | 3 (3) | 2 (2)
Angina pectoris (Cardiac disorders) | 5 (5) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT02742103/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT02742103/SAP_001.pdf